CLINICAL TRIAL: NCT05227547
Title: Mapping and Characterization of Alveolar Cells During Smoking and Chronic Obstructive Disease
Acronym: CoStemCells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Henri Mondor University Hospital (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CoStemCells
Record Dates: First submitted 2021-11-04; First posted 2022-02-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic resection surgery (Other): Smokers (active or ex-smokers) and non-smokers with COPD and without COPD undergoing thoracic resection surgery
  Interventions: Other: Thoracic resection surgery

INTERVENTIONS:
Other: Thoracic resection surgery — Patients undergoing thoracic resection surgery (pneumonectomy, lobectomy, segmentectomy) for cancer or suspected cancer, including smokers (active or ex-smokers) and non-smokers, with COPD and without COPD, and non-smoking patients.

SUMMARY:
To evaluate the regenerative capacities of mesenchymal cells composing the microenvironment of alveolar type 2 cells in a population of patients, undergoing thoracic surgery for suspected cancer, who are smokers with and without COPD compared to non-smokers patients

DETAILED DESCRIPTION:
Chronic obstructive pulmonary diseases (COPD) have a major public health impact, as evidenced by the 250 million patients affected by these diseases and the 50% 5-year mortality for severe stages of chronic obstructive pulmonary disease (COPD). One pathophysiological mechanism of COPD and emphysema is a depletion of alveolar progenitor cells inducing a loss of alveolar-reparation capacities after an aggression. The genesis of these alterations and the mechanisms involved remain unknown. Alveolar type 2 cells (AT2) are the alveolar epithelial progenitor cells. AT2 proliferate and differentiate into alveolar type 1 cells (AT1) which form the alveolar-capillary barrier, along with endothelial cells, through which respiratory gas exchanges take place. The proliferation and differentiation of AT2 into AT1 are under the control of mesenchymal cells and endothelial cells located in close proximity. Together these cells form the alveolar stem cell niche. The characteristics and interactions of the different cell populations have been well described during lung growth, in the normal adult lung or during pulmonary fibrosis; however, participants are poorly described during smoking exposure and chronic obstructive diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patient undergoing lung resection surgery (lobectomy, pneumonectomy, segmentectomy) for cancer or suspected cancer
3. Acceptance to participate in the protocol
4. Affiliated to a social security plan

Exclusion Criteria:

1. Chronic autoimmune disease
2. Patient under guardianship or curators
3. Neo-adjuvant chemotherapy
4. History of thoracic radiotherapy
5. Pregnant woman
6. Minor patient
7. Person not able to consent
8. Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2030-10-05 (Estimated); Study Completion 2030-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of alveolar organoids | through study completion, an average of 3 years
  Comparison of the number of alveolar organoids formed 21 days after culture of fibroblasts with alveolar type II cells between smokers with and without COPD and non-smoking patients

SECONDARY OUTCOMES:
Fibroblast proliferation capacity | through study completion, an average of 3 years
  Evaluated by their doubling time, number of cells collected compared to the number of cells seeded
Differentiation into myofibroblasts | through study completion, an average of 3 years
  By immunofluorescence marking: number of alpha-smooth muscle actin (alpha-SMA) + cells compared to total cells
Fibroblast migration capacity | through study completion, an average of 3 years
  Evaluated in Boyden chamber
Modulated signaling pathways in isolated fibroblasts between groups | through study completion, an average of 3 years
  Evaluated by Ribonucleic acid (RNA) sequencing of fibroblasts
Modulated signaling pathways in endothelial cells between groups | through study completion, an average of 3 years
  Evaluated byRibonucleic acid (RNA) sequencing of endothelial cells
Evaluation of cytokines in fibroblasts supernatant | through study completion, an average of 3 years
  Evaluated by Luminex Assay
Tumor progression | through study completion, an average of 3 years
  By studying the migration and invasion of tumor cells
Identification of different cell types on total lung | through study completion, an average of 3 years
  Cell types composing the lung stem cell microenvironment measured by single cell analysis
Severity of pulmonary emphysema, | At inclusion, every year, up to 5 years after surgery
  Change of lung density assessed by computed tomography scan
Type of pulmonary emphysema | At inclusion, every year, up to 5 years after surgery
  Assessed by computed tomography scan :
  [centro-lobular or pan-lobular, para-septal]
Research of pulmonary biomarkers | through study completion, an average of 3 years
  Searched according to the results obtained during cell cultures (immunohistochemistry, immunofluorescence)
Identification of biomarkers in the pre and postoperative circulating blood | through study completion, an average of 3 years
  Evaluated in laboratory by metagenomic analysis of 16s Ribonucleic acid (RNA) of bacteria for cluster analysis that correlate with lung injury and could be prognostic markers
Identification of biomarkers in the intestinal microbiota | through study completion, an average of 3 years
  Evaluated in laboratory by metagenomic analysis of 16s Ribonucleic acid (RNA) of bacteria for cluster analysis that correlate with lung injury and could be prognostic markers
Measurement of Forced expiratory volume at one second (FEV1) | through study completion, an average of 3 years
  Determine the relationship between respiratory disease phenotype and exercise impact by measurement of Forced expiratory volume at one second (FEV1)
Measurement of Forced Vital Capacity (FVC ) | through study completion, an average of 3 years
  Determine the relationship between respiratory disease phenotype and exercise impact by measurement of Forced Vital Capacity (FVC )
Measurement of pulmonary diffusion capacity of CO (DLCO) | through study completion, an average of 3 years
  Determine the relationship between respiratory disease phenotype and exercise impact by measurement of pulmonary diffusion capacity of CO (DLCO)
Measurement of CO transfer coefficient (KCO) | through study completion, an average of 3 years
  Determine the relationship between respiratory disease phenotype and exercise impact by measurement of CO transfer coefficient (KCO)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Rousseau-Bussac, Créteil
  - Hopital Cochin, Paris
  - HEGP, Paris
  - Hopital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No